CLINICAL TRIAL: NCT02968706
Title: High Flow Nasal Cannula Versus Conventional Nasal Cannula in Oxygen Performance in Patients Receiving Colonoscopy Under Intravenous Sedation
Brief Title: HFNC Versus Conventional Nasal Cannula in Oxygen Performance in Patients Receiving Colonoscopy Under IV Sedation
Acronym: HFNC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aventura Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-516
Record Dates: First submitted 2016-11-08; First posted 2016-11-21 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Desaturation of Blood
Keywords: High Flow Nasal Cannula; Colonoscopy; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High flow cannula arm (Experimental): Patients in the experimental arm (the high flow nasal cannula group) will receive heated humidified high flow oxygen of 50L/min at FiO2 of 40% throughout the colonoscopy. A patient satisfaction survey will be administered after procedure.
  Interventions: Device: High Flow Nasal Cannula; Other: Patient satisfaction questionnaire
- Conventional cannula arm (Active Comparator): Participants in control arm (the conventional nasal cannula group) will receive an oxygen flow of 2-5 L /min. A patient satisfaction survey will be administered after procedure.
  Interventions: Device: Conventional Nasal Cannula; Other: Patient satisfaction questionnaire

INTERVENTIONS:
Device: High Flow Nasal Cannula — Heated humidified high flow oxygen of 50 L/min at FiO2 of 40%
  Other Names: High flow oxygen delivering device (OPTIFLO)
  Arms: High flow cannula arm
Device: Conventional Nasal Cannula — Supplemental oxygen of 2-5 L/min
  Arms: Conventional cannula arm
Other: Patient satisfaction questionnaire — Questionnaire

SUMMARY:
The purpose of this study is to investigate if high flow nasal cannula (HFNC), as compared to conventional nasal cannula, improves oxygenation and prevents desaturation events in obese patients undergoing colonoscopy.

DETAILED DESCRIPTION:
Intravenous sedation during colonoscopy has become the standard practice in United States given its higher patient satisfaction and procedural quality. The most common used short acting sedative agent is propofol. Although possessing safe and rapidly reversed pharmacokinetic properties, propofol intravenous infusion can lead to respiratory depression and hypoxemia. In one prospective study, hypoxemia events, defined by oxygen saturation less than 90 percent was found in 20 percent of patients receiving colonoscopy using propofol sedation. The mechanism of hypoxemia is mainly hypoventilation, airway collapse, and carbon dioxide (CO2) retention. When it comes to gastrointestinal procedures, using oxygen devices for augmenting ventilation is usually avoided, ex: positive pressure ventilation, since it can lead to bowel distention and affect quality of procedures. Therefore most hospitals in United States still use nasal cannula of oxygen therapy during gastrointestinal procedures, and there is lack of available options of oxygen therapy which can improve hypoventilation and prevent hypoxemia.

High flow nasal cannula (HFNC) is a new generation of oxygen therapy. It provides constant high flow oxygen delivery with heated and humidified air. Moreover, it has been studied that high velocity of airflow can create the effect of "positive end expiratory pressure" thus assist ventilation and work of breathing. Compared to conventional nasal cannula and face mask, HFNC has demonstrated superior performance in oxygenation, work of breathing and patient comfort in many studies. Since its invention, HFNC has been studied in post-cardiac surgery, post-extubation, bronchoscopy and dental procedures and all of them show equal to better oxygen performance in comparison of nasal cannula.

While capnographic monitoring has been studied to prevent hypoxemia during sedation, no studies have been done to evaluate the clinical utility of new generation oxygen therapy. Obesity is associated with increased frequency of sedation related complications especially hypoxemia during propofol mediated sedation for advanced endoscopic procedures. The Investigators hypothesized that HFNC may improve oxygen performance compared to conventional nasal cannula for obese patients receiving colonoscopy under intravenous sedation.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30.
* Age ≥ 18 years.
* ASA classification II and III.
* Scheduled for colonoscopy.
* Able to provide written informed consent.

Exclusion Criteria:

* Allergic to propofol and any of its contents.
* Baseline SpO2 less than 93%.
* Patients who require intubation for airway protection based on anesthesiologist discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of desaturation events during procedures (desaturation events are defined by either SpO2 drops more than 5% compared to baseline SpO2 OR SpO2<90% at any time of procedures) | Through out the colonoscopy procedure (after propofol induction to the end of colonoscopy)

SECONDARY OUTCOMES:
Incidence rate of carbon dioxide retention (end tidal CO2 more than 50 mmHg at any time of procedure) | Through out the colonoscopy procedure (after propofol induction to the end of colonoscopy)
Patients satisfaction level (patient comfort and mouth dryness assessed by a questionnaire with 4-scale questions) | One time point (15 minutes after the patient recovered from anesthesia sedation)
Respiratory rates before and after colonoscopy procedure, and highest respiratory rate during colonoscopy procedure. | Three time points (Before, through out, and within 5 minutes after the colonoscopy procedure)
Incidence rate of hypoxia rescue intervention events (e.g. jaw lift, anterior mandibular shifting, head elevation ) | Through out the colonoscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hilda Mahmoudi, MD, MPH, Principal Investigator — Aventura Hospital and Medical Center
Locations (1):
- Aventura Hospital and Medical Center, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No